CLINICAL TRIAL: NCT05789667
Title: Observational Study on Gender-based Impact on Safety and Efficacy of Lenvatinib in Patients With Radioiodine Refractory Differentiated Thyroid Cancer
Brief Title: Gender-based Impact on Safety and Efficacy of Lenvatinib in Patients With Differentiated Thyroid Cancer
Acronym: Gisel
Status: Recruiting | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: University of Turin, Italy (Other); University of Roma La Sapienza (Other); University of Siena (Other); University of Pisa (Other); Istituto Oncologico Veneto IRCCS (Other); University of Catania (Other); Istituto Auxologico Italiano (Other)
Responsible Party: Principal Investigator, Marialuisa Appetecchia, Professor, Regina Elena Cancer Institute
Other Study IDs: RS1316/20(2312)
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Differentiated Thyroid Cancer; Gender
MeSH Terms: conditions — Coitus | interventions — lenvatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Lenvatinib — Patients will be treated by lenvatinib as recommended by good clinical practice
  Other Names: lenvatinib mesilate; Lenvatinib Oral Capsule [Lenvima]

SUMMARY:
Lenvatinib is approved for the treatment of radioiodine refractory differentiated thyroid cancer. Despite gender can play a crucial role un in safety and efficacy of oncological product, little is know on gender difference in lenvatinb effacacy and safety in the context of radioiodine refractory differentiated thyroid cancer.

The primary objective of the study is to assess safety and toxicity profile in male and female patients in terms of dose reduction. The secondary objectives are to assess sex and gender difference in: the number and the incidence of adverse events; response rate according to RECIST criteria 1.1; progression free survival, overall survival and duration of response.

DETAILED DESCRIPTION:
Lenvatinib is an orally available potent inhibitor of the split-kinase family of transmembrane growth factor receptors including Flt-1/VEGFR-1 and KDR/VEGFR. Lenvatinib has been investigated in hepatocellular carcinoma and in RAI-resistant thyroid cancer (Phase III trials) and in other malignancies, showing high rates of activity. In RAI-resistant thyroid cancer, lenvatinib showed a remarkable response rate over placebo (65% vs 2), combined with a prolonged progression free survival (18.3 vs 3.6 months). It has been approved for the treatment of locally recurrent or metastatic, progressive RAI resistance-DTC in the United States, Europe, and Japan, based on the results from SELECT trial. Moreover, lenvatinib demonstrated a meaningful clinical activity (response rate 64.8% in treatment arm vs 1.5% in placebo arm, p<0.001;) significantly reducing the tumour burden, with a median maximum percentage change in tumour size of -42.9%. Response was mostly pronounced at the first assessment (median -24.7% at 8 weeks after randomization) but it has been observed even in the following months (-1.3% per month). Recently, the efficacy of lenvatinib was confirmed in specific patient population, such as elderly. Although the efficacy is remarkable toxic effects are considerable and not all patients have the same risk to benefit ratio from lenvatinib treatment. Results derived from controlled clinical trials are rarely replicable in the real-life because these trials are usually conducted in selected populations, in a highly controlled setting, optimized to show the effect of the drug.

In this context growing evidences are showing gender associated functions playing a role in cancer incidence, progression and response to therapy; gender disparities in toxicities and effectiveness of certain drugs used in the treatment of the most common cancer is already well known.The aim of the present study is to evaluate the safety and efficacy profile of Lenvatinib based on gender in patients with refractory iodine DTC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with refractory iodine DTC treated with lenvatinib
* Signed written informed consent

Exclusion Criteria:

- Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by radio-refractory iodine differentiated thyroid cancer
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-05-27 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Gender difference in Safety profile of lenvatinib treatment | 1 year
  Difference in lenvatinib dose reduction between male and female patients

SECONDARY OUTCOMES:
Gender difference in lenvatinib side effects incidence | 1 year
  Difference in number of lenvatinib side effects between male and female patients according to CTCAE 5.0
Gender difference in lenvatinib response rate | 1 year
  Difference in lenvatinib response rate (CR+PR) according to RECIST response evaluation criteria 1.1 in male and female patients.
Gender difference progression free survival and overall survival of patients treated with lenvatinib | 1 year
  Difference in progression free survival and overall survival of patients treated with lenvatinib in male and female patients.

CONTACTS AND LOCATIONS:
Overall Officials: Marialuisa Appetecchia, Prof, Principal Investigator — Regina Elena Cancer Institute
Locations (1):
- Regina Elena National Cancer Institute, Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes
Raw data will be published in open access database
Time Frame: At the end of the study
Access Criteria: Open access
URL: http://garr.it